CLINICAL TRIAL: NCT06454019
Title: Evaluating Impact of Outreach Nudges Among Individuals Losing Medicaid Coverage in California
Brief Title: Phone Outreach Nudges Among Individuals Losing Medicaid Coverage
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Covered California (Other Government)
Responsible Party: Principal Investigator, Marina Lovchikova, Senior Research Data Scientist, Covered California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SB260-OCC-2023
Record Dates: First submitted 2024-06-05; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Behavioral Economics; Health Insurance
Keywords: Health Insurance; ACA marketplace; Behavioral Economics; Nudge

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group without a phone call (Experimental): Control Group was assigned to receive no phone outreach
  Interventions: Behavioral: Standard Notice
- Treatment Group with a phone call (Experimental): Treatment group was assigned to receive a phone call from Covered California call center
  Interventions: Behavioral: Phone Outreach

INTERVENTIONS:
Behavioral: Phone Outreach — Phone outreach to individuals losing Medicaid and auto-enrolled into Covered California plan to nudge them to act
  Arms: Treatment Group with a phone call
Behavioral: Standard Notice — Standard notification letter without phone outreach to individuals losing Medicaid and auto-enrolled into Covered California plan to nudge them to act
  Arms: Control Group without a phone call

SUMMARY:
In May 2023, Covered California, California's ACA marketplace, implemented its automatic enrollment program for individuals losing Medicaid coverage, as defined by Senate Bill 260. If individuals are found eligible for subsidized marketplace coverage, individuals will be automatically enrolled in the lowest cost silver plan available to them, but individuals must still take action to confirm their plan or pay their first month's premium. To identify whether the phone outreach is the effective outreach strategy to increase take-up in this population, Covered California implemented this intervention. The results of this evaluation will inform operational and budgeting decisions.

ELIGIBILITY:
Inclusion Criteria:

* Lost Medi-Cal (California's Medicaid coverage) in July 2023-June 2024
* Auto-enrolled into lowest cost silver plan with Covered California as per Senate Bill 260 and have not opted-in (effectuated) into the coverage
* Have a valid phone number on the health insurance application
* Do not have a delegated agent to their case
* Still have Covered California Program eligibility, not reverted back to Medi-Cal coverage
* Have English or Spanish as preferred speaking language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60045 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Health Plan Effectuation | within 30 days from the start date of plan they are auto-enrolled into
  A binary indicator for whether a consumer is effectuated into (paid for, opt-in into) Covered California plan, either the plan assigned through the auto-enrollment process, or into another plan chosen by the consumer by the end of the month at which outreach was conducted

SECONDARY OUTCOMES:
Tenure with Covered California (measured in months) | measured 1-2 years after the intervention
  A length of tenure with Covered California plan within calendar year and/or beyond
Office visit | measured 1-2 years after the intervention
  A binary indicator for whether someone had an office visit during 1-2 years since the intervention
Prescriptions filled | measured 1-2 years after the intervention
  A binary indicator for whether someone had a prescription drug fill during 1-2 years since the intervention
Emergency Room Visit | measured 1-2 years after the intervention
  A binary indicator for whether someone had an emergency room visit during 1-2 years since the intervention
Hospital admission | 1-2 years before and after the intervention
  A binary indicator for whether someone had a hospital admission 1-2 years before and 1-2 years after the intervention
Out-of-pocket spending on healthcare services | measured 1-2 years after the intervention
  Total out-of-pocket spending for the 1-2 years since the intervention
Uninsured | measured 1-2 years after the intervention
  A binary indicator for whether someone self-reported being uninsured while filing their taxes

CONTACTS AND LOCATIONS:
Overall Officials: Emory Wolf, MPP, Principal Investigator — Covered California
Locations (1):
- Covered California, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers are committed to sharing as much data as possible for replication, consistent with the privacy and security requirements of the state agency that govern the re-disclosure of the data.
Supporting Information: SAP
Time Frame: Data will be available with investigator support upon publication
Access Criteria: Replication data can be accessed via request to the primary investigator upon publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT06454019/Prot_SAP_000.pdf